CLINICAL TRIAL: NCT06514378
Title: An Open Label, Randomised, Controlled Clinical Trial to Asses the Safety of Endobronchial Administration of Allogneic Mesenchymal Stromal Cells in Patients With Lung Trasplant Chronic Rejection: Endosclad Study.
Brief Title: Safety of Endobronchial Mesenchymal Stromal Cells in the Treatment of Chronic Lung Allograft Dysfunction
Acronym: ENDOSCLAD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Instituto De Investigación Sanitaria Puerta De Hierro-Segovia De Arana (Other)
Collaborators: Ministerio de Ciencia, Innovación y Universidades (Unknown)
Responsible Party: Principal Investigator, David Gomez de Antonio, Head of Research Group, Instituto De Investigación Sanitaria Puerta De Hierro-Segovia De Arana
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICI/00122
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Chronic Lung Disease; Lung Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Biological: Mesenchymal stem cells
- Control (No Intervention)

INTERVENTIONS:
Biological: Mesenchymal stem cells — Endobronchial administration of 10⁶ MSCs/kg in each transplanted lung, 4 weeks apart.
  Arms: Treatment group

SUMMARY:
Lung transplantation is the only therapeutic alternative for more and more patients with respiratory diseases in their most advanced stages.

The most limiting factor to achieve long term survival si chronic lung allograft dysfunction, a multifactorial disease without an effective treatment.

The immunomodulatory capacity of mesenchymal stem cells enables them to be a potential therapeutic agent for this condition.

The objective of this study is to assess the safety of endobronchial administration of allogeneic MSCs in patients with chroniclung allograft dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Patients should have signed written informed consent. Adult patients ≥18 years of age at the time of enrolment Patients recipients of a uni or bipulmonary transplant An established diagnosis of BOS ≧ 0p (FEV1≤90% and / or FEF 25-75% ≤ of the baseline value with no other justifying cause) in the last 6 months.

Exclusion Criteria:

* History of lobar transplantation History of heart-lung transplantation Active infection at the time of inclusion. Active Acute Rejection not treated at the time of inclusion. Oncological history (except cutaneous basal cell or carcinoma in situ) Systemic autoimmune diseases. Active HIV / HBV / HCV infection (confirmed by serology or PCR) Proximal airway stenosis Pregnancy Performance status 3 or 4 (confined to bed or chair for more than 50% of waking hours, able only to perform some self-care activities) Estimated survival less than 3 months. Known hypersensitivity to components used in the production of allogeneic MSCs. Any circumstance that, in the opinion of the investigator, compromises the patient's ability to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Early onset adverse events | 24 hours
  Incidence of early onset (24h) adverse events following MSCs administration: desaturation, hypotension, radiological infiltrates, fever or changes in oxygen therapy requirements.
Adverse events | One year since randomization
  Incidence of adverse events of special interest since randomization: lower respiratory tract infections, acute rejection (as defined by the presence of A1-A4 o B1R, B2R in biopsy), BO worsening (as measured by >10% decline in FEV1 from baseline).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Puerta de Hierro Majadahonda, Madrid, Spain